CLINICAL TRIAL: NCT06667154
Title: Efficacy Analysis of Neoadjuvant Treatment in Lung Cancer Using Low-Dose Nivolumab Combined With Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aline Fusco Fares, MD (Other)
Collaborators: Hospital de Base de Sao Jose do Rio Preto (Unknown)
Responsible Party: Sponsor-Investigator, Aline Fusco Fares, MD, MD, Fundação Faculdade Regional de Medicina de São José do Rio Preto
Organization: Fundação Faculdade Regional de Medicina de São José do Rio Preto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungCancerLowDose
Record Dates: First submitted 2024-06-06; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer, Nonsmall Cell; Non-Small Cell Lung Cancer NSCLC
Keywords: Low Dose Immunotherapy; Neoadjuvant immunotherapy; Non-Small-Cell-Lung-Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low-dose nivolumab combined with platinum-based doublet chemotherapy (Experimental)
  Interventions: Drug: Low-dose nivolumab combined with platinum-based doublet chemotherapy

INTERVENTIONS:
Drug: Low-dose nivolumab combined with platinum-based doublet chemotherapy — Platinum-based neoadjuvant chemotherapy (carboplatin at AUC 5 or 6 combined with either paclitaxel at 175 mg/m² or pemetrexed at 500 mg/m²), administered with nivolumab at 0.3 mg/kg every 21 days for 3 cycles.

SUMMARY:
The primary objective of this study is to assess the major pathological response (MPR) rate and pathologic complete response (pCR) rate in stage IB-IIIA non-small cell lung cancer (NSCLC) treated with a low dose of neoadjuvant immunotherapy combined with platinum doublet.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide a signed Informed Consent Form (ICF), indicating agreement to comply with the requirements and restrictions in the ICF and protocol.
* Male or female, aged 18 years or older.
* Diagnosed with non-small cell lung cancer (NSCLC) with clinical staging IB, II, or IIIA.
* Receiving treatment at Hospital de Base.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment, with no decline from two weeks prior to the baseline period or the day of the first dose.
* Tumor sample meets the following requirements:
* Negative for EGFR gene expression.
* Negative for ALK and ROS1 protein expression.
* PD-L1 protein expression documented and assessable.
* Tumor is considered resectable upon initial assessment by three thoracic oncology surgeons (IR, CM, and HN) following a multidisciplinary review.
* Adequate organ and bone marrow function as defined below:
* Hemoglobin: ≥ 9.0 g/dL*
* Absolute neutrophil count: ≥ 1.5 × 10^9 /L*
* Platelet count: ≥ 100 × 10^9 /L*
* *Note: Granulocyte colony-stimulating factor (G-CSF), platelet transfusions, and blood transfusions are not permitted to meet these values.
* Serum bilirubin: ≤ 1.5 × upper limit of normal (ULN), except for participants with confirmed Gilbert syndrome, who may be included upon physician consultation.
* ALT and AST: ≤ 2.5 × ULN.
* Creatinine clearance: ≥ 50 mL/min (calculated using the Cockcroft and Gault formula).
* Life expectancy greater than six months prior to randomization.

Exclusion Criteria:

* Refusal to sign the Informed Consent Form (ICF).
* NSCLC clinical stages IA, IIIB N3, IIIC, IVA, and IVB.
* Tumors with T4 invasion of the aorta, esophagus, and/or heart; or presence of bulky N2 disease.
* Tumor deemed unresectable.
* Prior systemic anticancer therapy for NSCLC, including chemotherapy, biologic therapy, immunotherapy, or any investigational drugs.
* History of another primary malignancy, with exceptions for:
* Malignancies treated with curative intent and no active disease for ≥ 2 years before the first dose of investigational product (IP) and with a low risk of recurrence.
* Adequately treated non-melanoma skin cancer or lentigo maligna with no evidence of disease.
* Adequately treated carcinoma in situ with no evidence of disease.
* Incomplete basic medical information in the electronic medical record.
* Positive for EGFR gene expression.
* Positive for ALK protein expression.
* No available data on PD-L1 protein expression.
* Positive for ROS1 protein expression.
* Pregnant or breastfeeding at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response | 2-3 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
Pathologic Complete Response | 2-3 months
  Pathological complete response (pCR) is defined as having no residual cancer at the primary site or in regional lymph nodes on pathologic review of the surgical specimen.

SECONDARY OUTCOMES:
Adverse Events | Up to 3 months after the end of treatment
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.
Event-Free-Survival | Up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death.
R0 resection | Up to 3 months
  R0 resection rate is defined as the proportion of participants who have achieved R0 resection (complete resection with no residual tumor cell in the resection margin) in all participants.

OTHER OUTCOMES:
Rate of conversion from minimally invasive surgery to open surgery | 2-3 months
  The frequency at which a minimally invasive procedure needs to be converted to an open surgical approach mid-operation

CONTACTS AND LOCATIONS:
Overall Officials: JOAO A SOLER, MD, Principal Investigator — FUNDACAO FACULDADE REGIONAL DE MEDICINA DE SAO JOSE DO RIO PRETO
Locations (1):
- Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes